CLINICAL TRIAL: NCT01347723
Title: Scrambler Therapy for the Treatment of Chemotherapy Induced Peripheral Neuropathy: An Open Access Trial
Brief Title: Scrambler Therapy in Treating Pain and Peripheral Neuropathy in Patients Previously Treated With Chemotherapy
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC10CC; NCI-2011-00339 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC10CC (Other: Mayo Clinic Cancer Center); 11-000675 (Other: Mayo Clinic IRB); NCI-2011-00339 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-03-30; First posted 2011-05-04 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2016-01

CONDITIONS: Pain; Peripheral Neuropathy
MeSH Terms: conditions — Pain; Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Supportive care (pain therapy): Patients undergo scrambler therapy for 30 minutes daily for up to 10 consecutive days. Treatment continues in the absence of unacceptable toxicity.
  Interventions: Other: scrambler therapy; Other: questionnaire administration; Procedure: management of therapy complications

INTERVENTIONS:
Other: scrambler therapy — Undergo scrambler therapy
Other: questionnaire administration — Ancillary studies
Procedure: management of therapy complications — Undergo scrambler therapy
  Other Names: complications of therapy, management of

SUMMARY:
This pilot clinical trial studies scrambler therapy in treating pain and peripheral neuropathy in patients previously treated with chemotherapy. Scrambler therapy may help relieve pain from peripheral neuropathy caused by chemotherapy

DETAILED DESCRIPTION:
OBJECTIVES:

I. To record the types of patients that we treat, along with the reported efficacy and potential toxicity associated with scrambler therapy.

II. To get experience with patient reported outcome measurement tools that we use in this trial, including a report of analgesic use.

OUTLINE: Patients undergo scrambler therapy for 30 minutes daily for up to 10 consecutive days. Treatment continues in the absence of unacceptable toxicity. After completion of study treatment, patients are followed up for 10 weeks.

III. To explore neurologic testing changes in patients receiving scrambler therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pain or symptoms of neuropathy or pain of >= 1 month (30 days) duration for which the patient wants intervention
* Participants have to relate that tingling or pain was at least a four out of ten problem during the prior week, on a 0-10 scale where zero was no problem and ten was the worst possible problem and expected to have tingling or pain of at least 4/10 at the time of the first treatment
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) = 0, 1, or 2
* Life expectancy >= 3 months (90 days)
* Case review by the study chair, or designate, as a case where treatment should be tried.
* Ability to complete questionnaire(s) by themselves or with assistance - Ability to provide informed written consent

Exclusion Criteria:

* Pregnant women
* Patients with implantable drug delivery systems, e.g. Medtronic Synchromed
* Patients with heart stents or metal implants such as pacemakers, automatic defibrillators, aneurysm clips, vena cava clips and skull plates; (metal implants for orthopedic repair, e.g. pins, clips, plates, cages, joint replacements are allowed as are central venous access devices)
* Patients with a history of myocardial infarction or ischemic heart disease within the past six months
* Patients with history of epilepsy, brain damage, use of anti-convulsants for seizure prevention, concurrently using ketamine, symptomatic brain metastases; Note: anti-convulsant use is allowed for neuropathy and heart failure (HF) if on a stable dose
* Skin conditions such as open sores that would prevent proper application of the electrodes
* Other medical or other condition(s) that in the opinion of the investigators might compromise the objectives of the study
* Currently on gabapentin or pregabalin Note: (because of data that support that patients don't do as well when on gabapentin or pregabalin, all patients on these medications will be weaned off of them prior to study initiation. The study team will provide instructions on how to do this).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2011-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in pain on a 0-10 numerical rating scale. | 3 years

SECONDARY OUTCOMES:
Changes in neurologic function will be done by Neurometer Current Perception Threshold (CPT) testing and with a Rydel-Seiffer graduated tuning fork. | 3 years
  Patients will also undergo neurologic function testing. This will be done in an exploratory measure to try to correlate changes in the patient reported outcome instrument data with changes in the different measures of neurologic function. The two measures will be Neurometer Current Perception Threshold (CPT) Testing and testing with a Rydel-Seiffer graduated tuning fork.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Loprinzi, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States